CLINICAL TRIAL: NCT03465709
Title: An 18-Month Phase Ib/II Multi-Center, Open Label Study to Evaluate the Safety of Intravitreal APL-2 Therapy in Patients With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Pegcetacoplan (APL-2) in Neovascular AMD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Apellis concluded that sufficient data were collected to meet the study objectives.
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-203
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegcetacoplan Study Drug (Experimental)
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Study Drug
  Other Names: APL-2

SUMMARY:
Safety Assessment of Pegcetacoplan in Patients with Neovascular AMD

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 60 years.
2. Normal Luminance best corrected visual acuity (NL-BCVA) of 24 letters or better using Early Treatment Diabetic Retinopathy Study (ETDRS) charts (20/320 Snellen equivalent).
3. Clinical diagnosis of neovascular AMD with the following criteria met:

   1. Eligible for an injection of an anti-VEGF injection with macular fluid present at Day -28.
   2. Must have been treated with anti-VEGF in study eye for at least 6 months prior to joining the study.
   3. At least 6 months of intravitreal anti-VEGF therapy at intervals not greater than 8 weeks (± 7 days) for the past 2 injections in the eye that is selected to be the study eye.
4. A clinically meaningful (50%) reduction in excess macular fluid or macular thickness in the study eye at the discretion of the investigator between Screening Day -28 and Screening Day -14 as assessed by SD-OCT.
5. Female subjects must be:

   1. Women of non-child-bearing potential (WONCBP), or
   2. Women of child-bearing potential (WOCBP) with a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study and refrain from breastfeeding for the duration of the study.
6. Males with female partners of child-bearing potential must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study.
7. Willing and able to give informed consent and to comply with the study procedures and assessments

Exclusion Criteria:

1. Presence of other causes of choroidal neovascularization (CNV) including pathologic myopia (spherical equivalent ≥ -6 diopters), central serous chorioretinopathy, ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis.
2. History of vitrectomy to the study eye
3. Presence of any ophthalmologic condition that reduces the clarity of the media and that, in the opinion of the Investigator, interferes with ophthalmologic examination (e.g. advanced cataract or corneal abnormalities).
4. Intraocular surgery (including lens replacement surgery) within 3 months prior to randomization.
5. Any history of endophthalmitis.
6. Trabeculectomy or aqueous shunt or valve in the study eye.
7. Aphakia or absence of the posterior capsule. Note: previous violation of the posterior capsule is also excluded unless it occurred as a result of yttrium aluminum garnet (YAG) laser posterior capsulotomy in association with prior posterior chamber intraocular lens implantation and at least 60 days prior to baseline.
8. Any ophthalmic condition that may require surgery or medical intervention during the study period or, in the opinion of the Investigator, could compromise visual function during the study period (e.g. severe uncontrolled glaucoma, clinically significant diabetic macular edema, ischemic optic neuropathy, retinal vasculopathies).
9. Any contraindication to IVT injection including current ocular or periocular infection.
10. Current treatment for active systemic or localized infection.
11. Participation in any systemic experimental treatment or any other systemic investigational new drug within 6 weeks or 5 half-lives of the active (whichever is longer) prior to the start of study treatment. Note: clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary
12. Medical or psychiatric conditions that, in the opinion of the investigator, make consistent follow-up over the 24- month treatment period unlikely, or would make the subject an unsafe study candidate.
13. Any baseline laboratory value (hematology, serum chemistry or urinalysis) that in the opinion of the Investigator is clinically significant and not suitable for study participation.
14. Known hypersensitivity to fluorescein sodium for injection or hypersensitivity to pegcetacoplan or any of the excipients in pegcetacoplan solution

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Grossi, MD, PhD, Study Director — Apellis Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Apellis Clinical Site, Beverly Hills, California
  - Apellis Clinical Site, Hagerstown, Maryland
  - Apellis Clinical Site, Cleveland, Ohio
  - Apellis Clinical Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female subjects aged at least 60 years with a clinical diagnosis of neovascular age-related macular degeneration in the study eye were recruited to this Phase 1b/2, open-label study at 3 study centers in the United States conducted from 14 February 2018 until the last subject last visit on 05 April 2019.
Pre-assignment Details: Subjects who demonstrated a reduction in excess macular fluid or macular thickness based on spectral domain optical coherence tomography (SD-OCT) comparison between Screening Visits 1 and 2, and who were eligible received a first anti-vascular endothelial growth factor (anti-VEGF) injection at Visit 2 and a second one at baseline (Day 1, Visit 3).
Groups:
- 15 mg Pegcetacoplan: Intravitreal (IVT) injections of 15 milligrams (mg) pegcetacoplan once monthly for 12 months, followed by a 6-month safety follow-up period.
Period: Overall Study
Arm/Group | 15 mg Pegcetacoplan
Started (Received at least 1 dose pegcetacoplan.) | 17
Completed (Completed planned treatment phase to Visit 15.) | 0
Not Completed | 17
Not completed — Study/Site Terminated by Sponsor | 14
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: The safety set included all subjects who received at least 1 dose of pegcetacoplan.
Groups:
- 15 mg Pegcetacoplan: IVT injections of 15 mg pegcetacoplan once monthly for 12 months, followed by a 6-month safety follow-up period.
Arm/Group | 15 mg Pegcetacoplan
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Native Hawaiian or Other Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Ocular and Systemic Treatment-Emergent Adverse Events (TEAEs) Including by Maximum Severity
Description: TEAEs were defined as those adverse events (AEs) that developed or worsened after the first dose of study drug, up to 30 days after the last dose. The severity of the TEAEs was classified as mild (asymptomatic/mild symptoms); moderate (minimal, local/non-invasive intervention indicated); severe (medically significant but not life-threatening); life-threatening or leading to death. The number of subjects experiencing 1 TEAE in each category is presented. A maximum of 7 injections of pegcetacoplan (per subject) and a maximum of 13 injections of anti-VEGF (per subject) were received during the study.
Time Frame: Day 1 up to end of study (up to 1 year).
Population: The safety set included all subjects who received at least 1 dose of pegcetacoplan.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg Pegcetacoplan
Number analyzed (Participants) | 17
Participants
  Any TEAEs | 15
  Ocular study eye TEAE | 14
  Nonocular TEAE | 7
  TEAE at least possibly related to study drug | 5
  TEAE at least possibly related to injection | 8
  Serious TEAEs | 4
  TEAEs leading to study drug discontinuation | 1
  TEAEs leading to death | 0
  Maximum severity: mild | 6
  Maximum severity: moderate | 6
  Maximum severity: severe | 3
  Maximum severity: life-threatening | 0

2. Secondary Outcome: Mean Change From Baseline in SD-OCT Central Subfield Thickness (CST) up to 12 Months
Description: The CST was measured using SD-OCT throughout the study and the mean change from baseline at each timepoint is presented for the study eye.
Time Frame: Day 1 up to Day 360 (12 months).
Population: The intent-to-treat set included all subjects who received at least 1 dose of pegcetacoplan.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | 15 mg Pegcetacoplan
Number analyzed (Participants) | 17
micrometers
  Day 30 | 12.9 (39.06)
  Day 60: number analyzed (Participants) | 15
  Day 60 | 16.1 (66.99)
  Day 90: number analyzed (Participants) | 16
  Day 90 | 15.1 (57.44)
  Day 120: number analyzed (Participants) | 15
  Day 120 | 31.6 (68.33)
  Day 150: number analyzed (Participants) | 15
  Day 150 | 34.8 (90.50)
  Day 180: number analyzed (Participants) | 15
  Day 180 | 48.3 (92.21)
  Day 210: number analyzed (Participants) | 15
  Day 210 | 18.5 (66.06)
  Day 240: number analyzed (Participants) | 15
  Day 240 | 34.1 (66.35)
  Day 270: number analyzed (Participants) | 15
  Day 270 | 49.2 (58.76)
  Day 300: number analyzed (Participants) | 13
  Day 300 | 22.2 (73.29)
  Day 330: number analyzed (Participants) | 10
  Day 330 | -0.7 (57.17)
  Day 360: number analyzed (Participants) | 4
  Day 360 | -10.5 (48.67)

3. Secondary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Physical Examination Findings, Vital Signs and Laboratory Parameters
Description: Physical examinations, vital signs and laboratory parameters were monitored throughout the study and any subjects showing a clinically significant change from baseline over the study period are presented.
Time Frame: Baseline (Screening or Day 1) up to end of study (up to 1 year).
Population: The safety set included all subjects who received at least 1 dose of pegcetacoplan.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg Pegcetacoplan
Number analyzed (Participants) | 17
Participants
  Physical examination findings | 2
  Vital signs | 0
  Laboratory parameters | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to end of study (up to 1 year).
Description: The safety set included all subjects who received at least 1 dose of pegcetacoplan. Ocular TEAEs are presented separately for the study and fellow eyes, and non-ocular (systemic) TEAEs are also presented.
Groups:
- 15 mg Pegcetacoplan: Ocular Study Eye: Ocular TEAEs are summarized for the study eye for all subjects who received IVT injections of 15 mg pegcetacoplan once monthly for 12 months.
- 15 mg Pegcetacoplan: Ocular Fellow Eye: Ocular TEAEs are summarized for the fellow eye for all subjects who received IVT injections of 15 mg pegcetacoplan once monthly for 12 months.
- 15 mg Pecgectacoplan: Non-ocular: Non-ocular (systemic) TEAEs are summarized for all subjects who received IVT injections of 15 mg pegcetacoplan once monthly for 12 months.
Arm/Group | 15 mg Pegcetacoplan: Ocular Study Eye | 15 mg Pegcetacoplan: Ocular Fellow Eye | 15 mg Pecgectacoplan: Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 3/17 | 0/17 | 1/17
Other Adverse Events (participants affected / at risk) | 13/17 | 3/17 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Pegcetacoplan: Ocular Study Eye (N=17) | 15 mg Pegcetacoplan: Ocular Fellow Eye (N=17) | 15 mg Pecgectacoplan: Non-ocular (N=17)
Uveitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Non-infectious endophthalmitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Pegcetacoplan: Ocular Study Eye (N=17) | 15 mg Pegcetacoplan: Ocular Fellow Eye (N=17) | 15 mg Pecgectacoplan: Non-ocular (N=17)
Uveitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (4) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 5 (8) | 0 (0) | 0 (0)
Optic nerve cup/disc ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitiviy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Exposure was shorter than expected as some subjects experienced intraocular inflammation in the study eye due to an identified impurity. The sponsor terminated the study early as sufficient data were collected to meet study objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT03465709/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT03465709/SAP_001.pdf